CLINICAL TRIAL: NCT05376540
Title: Norwegian Randomized Trial on Indocyanine Green Cholangiography Utility for Laparoscopic Cholecystectomy, Prestudy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REK280193
Record Dates: First submitted 2022-01-27; First posted 2022-05-17 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Gall Stone; Cholecystitis
Keywords: Cholecystectomy; Flourescent cholangiography
MeSH Terms: conditions — Gallstones; Cholecystitis | interventions — Injections, Intravenous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Direct gallbladder injection (Other): 2.5 mg of ICG will be injected directly into gallbladder intraoperatively.
  Interventions: Procedure: Direct gallbladder injection of ICG intraoperatively
- 2.5 mg intravenously (Other): 2.5 mg will ICG will be injected intravenously 1 hour prior to surgery.
  Interventions: Procedure: Intravenous injection 2.5 mg
- 2.5 mg intravenously + direct gallbladder injection (Other): 2.5 mg ICG will be injected intravenously 1 hour prior to surgery and another 2.5 mg ICG will be injected directly into the gallbladder intraoperatively.
  Interventions: Procedure: Intravenous injection and direct gallbladder injection
- 5 mg intravenously (Other): 5 mg ICG will be injected intravenously 0-8 hours prior to surgery.
  Interventions: Procedure: Intravenous injection 5 mg

INTERVENTIONS:
Procedure: Direct gallbladder injection of ICG intraoperatively — Patients randomized to this arm will have 2.5 mg ICG injected directly into the gallbladder intraoperatively.
  Arms: Direct gallbladder injection
Procedure: Intravenous injection 2.5 mg — Patients randomized to this arm will have 2.5 mg ICG injected intravenously 1 hour prio to surgery
  Arms: 2.5 mg intravenously
Procedure: Intravenous injection and direct gallbladder injection — Patients randomized to this arm will have 2.5 mg ICG injected intravenously 1 hour prior to surgery and another 2.5 mg ICG injected directly into the gallbladder, intraoperatively.
  Arms: 2.5 mg intravenously + direct gallbladder injection
Procedure: Intravenous injection 5 mg — Patients randomized to this arm will have 5 mg ICG injected intravenously 0-8 hours prior to surgery
  Arms: 5 mg intravenously

SUMMARY:
The purpose of this study is to compare different dosages and ways of administration of indocyanine green during fluorescent cholangiography in laparoscopic cholecystectomy. The study is randomized.

ELIGIBILITY:
Inclusion Criteria:

* Indication for laparoscopic cholecystectomy
* Signed informed consent

Exclusion Criteria:

* Allergy to indocyanine green or iodine
* Pregnancy or breast feeding

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
A questionnaire will be used to evaluate the surgeons experience. | 3-4 months
  This study aims to compare the surgeons subjective experience of ICG utility for different dosages and route of administration of indocyanine green in patients operated with laparoscopic cholecystectomy. A questionnaire will be used to evaluate the surgeons experience.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Nordby, MD, PhD, Principal Investigator — Ostfold Hospital Trust, Norway
Locations (1):
- Østfold Hospital trust, Moss, Norway

IPD SHARING:
Plan to Share IPD: No